CLINICAL TRIAL: NCT00680758
Title: A Phase I Study of Cisplatin, Paclitaxel, and RAD001 Patients With Metastatic Breast Cancer
Brief Title: Cisplatin, Paclitaxel, and Everolimus in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0770; VU-VICC-BRE-0770
Record Dates: First submitted 2008-05-18; First posted 2008-05-20 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Cisplatin; Everolimus; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: cisplatin; Drug: everolimus; Drug: paclitaxel

INTERVENTIONS:
Drug: cisplatin — * Dose Level: -3 20mg/m2/week 3-6 patients
  * Dose Level: -2 20mg/m2/week 3-6 patients
  * Dose Level: -1 25mg/m2/week 3-6 patients
  * Dose Level: 1 25mg/m2/week 3-6 patients
  * Dose Level: 2 25mg/m2/week 3-6 patients
  * Dose Level: 3 25mg/m2/week 3-6 patients
  Other Names: Platinol
Drug: everolimus — * Dose Level: -3 20mg/m2/week 3-6 patients
  * Dose Level: -2 20mg/m2/week 3-6 patients
  * Dose Level: -1 20mg/m2/week 3-6 patients
  * Dose Level: 1 20mg/m2/week 3-6 patients
  * Dose Level: 2 25mg/m2/week 3-6 patients
  * Dose Level: 3 30mg/m2/week 3-6 patients
  Other Names: RAD001
Drug: paclitaxel — * Dose Level: -3 65mg/m2/week 3-6 patients
  * Dose Level: -2 70mg/m2/week 3-6 patients
  * Dose Level: -1 70mg/m2/week 3-6 patients
  * Dose Level: 1 80mg/m2/week 3-6 patients
  * Dose Level: 2 80mg/m2/week 3-6 patients
  * Dose Level: 3 80mg/m2/week 3-6 patients
  Other Names: Taxol

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving more than one drug (combination chemotherapy) together with everolimus may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of cisplatin, paclitaxel, and everolimus when given together for the treatment of patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the safety profile and the maximum tolerated dose of the combination of cisplatin, paclitaxel, and everolimus in patients with metastatic breast cancer.

Secondary

* To explore the antitumor activity of this regimen, in terms of response rate and time to progression in these patients.

OUTLINE: This is a multicenter study.

Patients receive cisplatin intravenously (IV) over 1 hour and paclitaxel IV over 1 hour on days 1, 8, and 15. Patients receive oral everolimus on days 1, 8, 15, and 21. Courses repeat every 4 weeks in the absence of disease progression and unaccepted toxicity.

After completion of study therapy, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed invasive mammary carcinoma

  * Stage IV disease
* No locally recurrent breast cancer
* Patients with HER2/neu overexpressing tumors must have received prior trastuzumab (Herceptin®) in first-line treatment of metastatic breast cancer
* Patients with estrogen receptor- or progesterone receptor-expressing tumors must have received prior endocrine therapy (i.e., aromatase inhibitors, fulvestrant, tamoxifen, or ovarian ablation) in first-line treatment of metastatic breast cancer
* No symptomatic brain metastases

  * Patients with a history of brain metastases must be clinically stable and not taking steroids or therapeutic anticonvulsants that are CYP3A4 modifiers
  * Patients with asymptomatic brain metastases on prophylactic convulsants that are CYP3A4 modifiers are not eligible
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* ANC ≥ 1000/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN (3 times ULN if liver metastasis present)
* SGOT and SGPT ≤ 1.5 times ULN (3 times ULN if liver metastasis present)
* Alkaline phosphatase ≤ 3 times ULN if liver metastasis present
* Able to swallow and retain oral medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Must be disease-free from prior invasive cancers for > 5 years with the exception of completely resected basal cell or squamous cell carcinoma of the skin or successfully treated cervical carcinoma in situ
* No malabsorption syndrome, disease significantly affecting gastrointestinal function, or ulcerative colitis
* No uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring parenteral antibiotics
  * Impairment of lung function (i.e., chronic obstructive pulmonary disease or lung conditions requiring oxygen therapy)
  * Symptomatic New York Heart Association class III-IV congestive heart failure
  * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within the past 6 months
  * Uncontrolled hypertension (systolic blood pressure [BP] > 180 mm Hg or diastolic BP > 100 mm Hg)
  * Clinically significant cardiac arrhythmia (i.e., multifocal premature ventricular contractions, bigeminy, trigeminy, or ventricular tachycardia that is symptomatic or requires treatment)
  * Uncontrolled diabetes
  * Psychiatric illness/social situations that would preclude compliance with study requirements
* No known history of uncontrolled or symptomatic neuropathy ≥ grade 2
* No hypersensitivity to paclitaxel, or drugs using the vehicle Cremophor, Chinese hamster ovary cell products, or other recombinant human antibodies

Exclusion Criteria:

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior treatment
* Must not have exceeded a total cumulative dose of life-time exposure of doxorubicin hydrochloride ≤ 360 mg/m² or epirubicin hydrochloride ≤ 640 mg/m²
* At least 2 weeks since other prior investigational drugs
* No prior resection of the stomach or small bowel
* No more than 4 prior chemotherapy regimens in the metastatic setting

  * This restriction does not include endocrine therapies or single agent biologic therapies (i.e., trastuzumab)
* Concurrent radiotherapy to painful bone metastases or areas of impending bone fracture allowed as long as radiotherapy is initiated prior to study entry
* No concurrent trastuzumab
* No concurrent endocrine therapy
* No concurrent CYP3A4 modifiers
* No concurrent herbal supplement
* No other concurrent anticancer therapy (chemotherapy, radiotherapy, surgery, immunotherapy, hormonal therapy, or biological therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety profile and maximum tolerated dose | At 4 weeks
  The Maximum Tolerated Dose (MTD) will be the dose level at which fewer than 2 of 6 (or 33% of) patients experience dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Antitumor activity | Date of study entry to date of progression of disease
  Cisplatin + Paclitaxel + RAD001 combination by determining response rates (RR) and time to progression (TTP) achieved with treatment
Response rate | at baseline and every 8 weeks to disease progression
Time to progression | date of study entry to date of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee